CLINICAL TRIAL: NCT04490343
Title: Detection of Urinary Tract Stones on Ultra-low Dose Abdominopelvic CT Imaging With Deep-learning Image Reconstruction Algorithm
Brief Title: Detection of Urinary Stones on ULDCT With Deep-learning Image Reconstruction Algorithm
Acronym: URO DLIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2020_843_0053
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Urolithiasis; Urinary Tract Stones; Renal Colic; Deep Learning Reconstruction
Keywords: Urolithiasis; Urinary Tract Stones; Renal Colic; deep learning reconstruction; radiation dose; dose reduction; low dose CT
MeSH Terms: conditions — Urolithiasis; Urinary Calculi; Renal Colic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Abdominopelvic low dose CT — Patients with urinary stones will undergo multiple computed tomography (CT) examinations

SUMMARY:
Urolithiasis has an increasing incidence and prevalence worldwide, and some patients may have multiple recurrences. Because these stone-related episodes may lead to multiple diagnostic examinations requiring ionizing radiation, urolithiasis is a natural target for dose reduction efforts. Abdominopelvic low dose CT, which has the highest sensitivity and specificity among available imaging modalities, is the most appropriate diagnostic exam for this pathology. The main objective of this study is to evaluate the diagnostic performance of ultra-low dose CT using deep learning-based reconstruction in urolithiasis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Patient referred for abdominopelvic CT to confirm urolithiasis or for follow-up,
* Affiliation to a social security program,
* Ability of the subject to understand and express opposition

Exclusion Criteria:

* Age <18 years old,
* Person under guardianship or curators,
* Pregnant woman,
* Any contraindications to CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy between low dose CT using DLIR reconstruction and low dose CT without DLIR reconstruction for the detection of urinary tract stones | day 1
  Accuracy between low dose CT using DLIR reconstruction and low dose CT without DLIR reconstruction for the detection of urinary tract stones.
  Patients who were referred to the department for abdominopelvic CT exam for urolithiasis diagnostic or follow-up, and had consented to participate in the study, will undergo an additional ultra-low dose acquisition (ULD, <1 mSv) with deep learning-based reconstruction (DLIR).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No